CLINICAL TRIAL: NCT03547362
Title: Real-time Amino Acid Profiling
Acronym: RAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NIZO Food Research (Other)
Collaborators: FrieslandCampina (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: NL65184.072.18
Record Dates: First submitted 2018-04-20; First posted 2018-06-06 (Actual); Last update posted 2018-07-11 (Actual); Status verified 2018-07

CONDITIONS: Protein Digestion Kinetics
Keywords: Amino acids; Dairy proteins; Postprandial; Older adults
MeSH Terms: interventions — Caseins; Whey Proteins

STUDY DESIGN:
Intervention Model Description: The study is designed as a randomized, single-blinded within-subject (cross-over) trial in which a group of 12 subjects receive 6 different dairy products.
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Casein (Experimental): Single oral administration
  Interventions: Dietary Supplement: Casein
- Dairy protein blend 1 (Experimental): single oral administration
  Interventions: Dietary Supplement: Dairy protein blend 1
- Whey protein (Experimental): Single oral administration
  Interventions: Dietary Supplement: Whey protein
- Dairy protein blend 2 (Experimental): Single oral administration
  Interventions: Dietary Supplement: Dairy protein blend 2
- Dairy protein blend 3 (Experimental): Single oral administration
  Interventions: Dietary Supplement: Dairy protein blend 3
- Dairy protein blend 4 (Experimental): Single oral administration
  Interventions: Dietary Supplement: Dairy protein blend 4

INTERVENTIONS:
Dietary Supplement: Casein — See arm description
  Arms: Casein
Dietary Supplement: Dairy protein blend 1 — See arm description
  Arms: Dairy protein blend 1
Dietary Supplement: Whey protein — See arm description
  Arms: Whey protein
Dietary Supplement: Dairy protein blend 2 — See arm description
  Arms: Dairy protein blend 2
Dietary Supplement: Dairy protein blend 3 — See arm description
  Arms: Dairy protein blend 3
Dietary Supplement: Dairy protein blend 4 — See arm description
  Arms: Dairy protein blend 4

SUMMARY:
This study was designed to obtain information about the effect of new combinations of dairy proteins, in small servings with high protein concentrations, on postprandial amino acid kinetics in blood in an older population.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥65 and ≤80
* BMI ≥20 and ≤32 kg/m2
* Non-smoking
* Healthy as assessed by the NIZO lifestyle and health questionnaire ("Verklaring leefgewoonten en gezondheid") and according to the judgment of the study physician.
* Regular and normal Dutch eating habits as assessed by the NIZO lifestyle and health questionnaire (3 main meals per day)
* Veins suitable for cannulation (blood sampling)
* Voluntary participation
* Having given written informed consent
* Willing to comply with study procedures
* Accept use of all encoded data, including publication, and the confidential use and storage of all data for 15 years.
* Accept disclosure of the financial benefit of participation in the study to the authorities concerned

Exclusion Criteria:

* Participation in any clinical trial including blood sampling and/or administration of substances up to 30 days before day 1 of this study
* Having a history of medical or surgical events that may significantly affect the study outcome, including: Inflammatory bowel disease, hepatitis, pancreatitis, ulcers, gastrointestinal or rectal bleeding; major gastrointestinal tract surgery such as gastrectomy, gastroenterostomy, or bowel resection; known or suspected gastrointestinal disorders, colon or GI tract cancer
* Use of the following medication: glucose lowering drugs, insulin; medication that may impact gastric emptying (e.g. gastric acid inhibitors or laxatives)
* Diagnosed with diabetes, being treated for high blood glucose or increased fasting blood glucose (> 7 mmol/l in finger prick blood) as assessed during screening visit
* For men: Hb <8,5 mmol/l as assessed during screening visit; for women: Hb <7,5 mmol/l.
* Use of protein supplements
* Mental status that is incompatible with the proper conduct of the study
* A self-reported reported food allergy or sensitivity to dairy ingredients
* Alcohol consumption for men > 28 units/week and >4/day; for women: >21 units/week and >3/day
* Reported unexpected weight loss or weight gain of > 3 kg in the month prior to pre-study screening, or intention to lose weight during the study period
* Reported slimming or medically prescribed diet
* Recent blood donation (<1 month prior to Day 01 of the study)
* Not willing to give up blood donation during the study
* Personnel of NIZO food research and FrieslandCampina, their partner and their first and second degree relatives
* Not having a general practitioner
* Not willing to accept information-transfer concerning participation in the study, or information regarding his or her health, like laboratory results and eventual adverse events to and from his general practitioner

Ages: 65 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2018-07-05 (Actual); Study Completion 2018-07-05 (Actual)

PRIMARY OUTCOMES:
Postprandial serum amino acid concentration | 0-300 min after consumption
  Blood amino acid concentrations (mmol/L) before and at 13 time points (up till 5 hours) after consumption of the dairy products.

CONTACTS AND LOCATIONS:
Overall Officials: Melle van Schaik, Study Director — NIZO Food Research
Locations (1):
- NIZO Food Research, Ede, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No